CLINICAL TRIAL: NCT00543751
Title: Placebo Controlled Metformin and Sulfonylurea Combination Study in Patients With Type 2 Diabetes (0767-025)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0767-025; 2007_634; MK-0767-025
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — MK0767

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0767

SUMMARY:
The purpose of this study is to compare how MK0767 and metformin and sulfonylurea therapy lower blood glucose in patients with inadequate glycemic control This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes wtih inadequate glycemic control on maximally effective/tolerated metformin and sulfonylurea therapy
* Non-pregnant females

Exclusion Criteria:

* Patients with Type 1 Diabetes or history of ketoacidosis
* Patients who have been treated with insulin or other antihyperglycemic agents
* Patients with viral hepatitis, active liver or gallbladder disease, history of pancreatitis, heart disease, congestive heart failure, inadequately controlled hypertension, HIV positive, history hematologic disorders or neoplastic disease

Ages: 21 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2003-01; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC